CLINICAL TRIAL: NCT04460326
Title: Comparison of Postprandial Glycemic Control in Non-critically Ill Hospitalized Patients With Type 2 Diabetes Mellitus Using Novolog vs. Fiasp Insulin: a Randomized Controlled Open Label Trial
Brief Title: Novolog vs. Fiasp Insulin in Non-critically Ill Hospitalized Patients With Type 2 Diabetes Mellitus
Acronym: In-FI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-39600
Record Dates: First submitted 2020-06-04; First posted 2020-07-07 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Type 2 Diabetes Treated With Insulin
Keywords: Fiasp; Novolog; Continuous glucose monitor (CGM); Hypoglycemia; Hyperglycemia; Hemoglobin A1c
MeSH Terms: conditions — Hypoglycemia; Hyperglycemia | interventions — Insulin Glargine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 insulin glargine and Novolog (Active Comparator): Group 1 will receive daily basal insulin glargine with a scheduled bolus of meal insulin Novolog. Meal Novolog will be dosed at the time the subject starts to eat. If the premeal blood glucose (BG) is ≥ 150 mg/dL, additional Novolog will be administered based off the correctional scale at the same time as the prandial insulin. The dose of Novolog will be administered by the floor nurse as per usual standard of care.
  Interventions: Drug: Insulin glargine; Drug: NovoLog; Other: Standard carbohydrate diet
- Group 2 insulin glargine and Fiasp (Experimental): Group 2 will receive basal insulin glargine as dosed in Group 1. Meal insulin Fiasp dosing will be calculated the same way as Novolog dosing. If the premeal BG is ≥ 150 mg/dL, additional Fiasp will be administered based off the correctional scale at the same time as the prandial insulin.
  Interventions: Drug: Insulin glargine; Drug: Insulin Fiasp; Other: Standard carbohydrate diet

INTERVENTIONS:
Drug: Insulin glargine — Insulin glargine doses will be determined by calculating the total daily dose (TDD) of insulin and providing 50% of the TDD as follows: start at 0.5 units/kg/day and subtract 0.1 unit/kg/day for 70+ yrs of age, renal insufficiency, pancreatic deficiency and add 0.1 unit/kg/day if hemoglobin A1c in >10%
  Other Names: Lantus®
Drug: NovoLog — Novolog will be administered with each meal if premeal glucose is ≥ 150 mg/dL and at bedtime if glucose is ≥ 200 mg/dL by calculating an individualized insulin sensitivity factor for each subject per the following formula: 1500/total daily dose of insulin = sensitivity factor.
  Other Names: NovoLog®
  Arms: Group 1 insulin glargine and Novolog
Drug: Insulin Fiasp — Fiasp will be administered with each meal if premeal glucose is ≥ 150 mg/dL and at bedtime if glucose is ≥ 200 mg/dL by calculating an individualized insulin sensitivity factor for each subject per the following formula: 1500/total daily dose of insulin = sensitivity factor.
  Other Names: Fiasp®
  Arms: Group 2 insulin glargine and Fiasp
Other: Standard carbohydrate diet — Standard carbohydrate diet as per usual hospital care (75g with each meal)

SUMMARY:
Hyperglycemia affects 30-40% of hospitalized patients. Despite the fact that basal/bolus insulin therapy has been demonstrated to improve glycemic control and clinical outcomes in patients, achieving good glucose control remains a challenge.

This study examines the effects of Fiasp (a faster acting insulin) on blood sugars after meals compared to another type of insulin known as Novolog. The study will be performed in patients with type 2 diabetes admitted to the hospital, who are not in the intensive care unit, and who are being seen by the inpatient diabetes consult team. Eligible participants will be treated with Fiasp or Novolog injected multiple times a day before meals and at bedtime, in addition to a once daily injection of insulin glargine as basal insulin. Which type of meal time insulin (Fiasp vs Novolog) the subject gets is decided by chance, like the flip of a coin. Insulin doses will be started and titrated based on a protocol. All the subjects will wear a blinded continuous glucose monitoring (CGM)) sensor placed in their arm which they will wear for 72 hours during the study. The glucose values from the CGM, collected during the time it is worn, will be downloaded and compared to assess the response to the two different types of insulins - Fiasp and Novolog. The goal is to determine if Fiasp works as well as or better than Novolog in controlling blood sugars, particularly after meals, in the subjects of the study.

ELIGIBILITY:
Inclusion criteria

1. English-speaking
2. Males and female adult subjects admitted to Boston Medical Center to a medical or surgical floor.
3. Consultation by the Inpatient Diabetes Service at Boston Medical Center is required prior to consent.
4. Age ≥ 21 and <= 80 years.
5. Diagnosed with type 2 diabetes at least 180 days prior to screening.
6. Hyperglycemia during admission, as defined by a point of care and/or venous blood glucose ≥ 140 mg/dL.
7. Prior to admission subjects must be using one of the following for outpatient diabetes management:

   1. Insulin
   2. ≥ 2 oral/injectable agents
   3. One oral/injectable agent with a hemoglobin A1c of ≥ 8% within 3 months of enrollment.
8. Patients who are expected to remain hospitalized for a minimum of 48 hours following CGM sensor placement.
9. BMI <45 kg/m^2.
10. Subjects must have insulin glargine dosing planned at bedtime for the duration of the study period. Morning and afternoon dosing of insulin glargine are exclusionary.

Exclusion criteria:

1. Patients with a history of type 1 diabetes or late-onset autoimmune diabetes (LADA).
2. Treatment or plan for treatment with glucocorticoids during the index hospitalization.
3. Female patients who are pregnant (tested during hospitalization or screening) or breast-feeding during the hospitalization.
4. Patients admitted with the following conditions: diabetic ketoacidosis, hyperosmolar hyperglycemic state, solid organ transplantation, or coronary artery bypass surgery.
5. Prior diagnosis of gastroparesis or cirrhosis.
6. Acute or chronic kidney disease with a serum creatinine of ≥ 2 mg/dL at the time of screening.
7. Clinically significant nausea and/or vomiting or unable to consume more than 30 grams of carbohydrate at each meal.
8. Patients expected to receive nothing by mouth (NPO) for >24 hours.
9. Use of continuous or intermittent enteral feeding or parenteral nutrition.
10. Patient receiving aspirin and/or vitamin C during the hospitalization.
11. Any mental condition rendering the subject unable to provide informed consent.
12. Patients currently incarcerated.
13. Patients using >1 unit/kg/day of insulin prior to admission.
14. Insulin pump usage within the 2 weeks prior to or during admission.
15. Patients currently using real-time continuous glucose monitoring (CGM) or personal flash glucose monitoring system (FGM).
16. Patients with a history of an allergy to any of the types of insulin or one of the excipients in the insulin used in the study.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2023-05-27 (Actual); Study Completion 2023-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara M Alexanian, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Completed at Least 4 Meals
Arm/Group | Group 1 Insulin Glargine and Novolog | Group 2 Insulin Glargine and Fiasp
Started | 68 | 69
Completed | 61 | 61
Not Completed | 7 | 8
Not completed — Early discharge | 5 | 5
Not completed — Started oral antihyperglycemic | 1 | 1
Not completed — Nutrition method changed | 1 | 0
Not completed — Transfer to ICU | 0 | 1
Not completed — Bleeding at CGM site | 0 | 1
Period: Insulin Boluses & Postprandial CGM Data
Arm/Group | Group 1 Insulin Glargine and Novolog | Group 2 Insulin Glargine and Fiasp
Started | 61 | 61
Completed | 56 | 49
Not Completed | 5 | 12
Not completed — Postprandial or CGM data not available | 5 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 Insulin Glargine and Novolog | Group 2 Insulin Glargine and Fiasp | Total
Number analyzed (Participants) | 68 | 69 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (12) | 59.4 (10.1) | 58 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 46
  Male | 44 | 47 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 20 | 42
  Not Hispanic or Latino | 45 | 49 | 94
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 35 | 33 | 68
  White | 21 | 20 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 16 | 27
Region of Enrollment [Number; unit: participants]
  United States | 68 | 69 | 137
Diabetes treatment prior to admission [Count of Participants; unit: Participants]
  Insulin use | 45 | 43 | 88
  Non-insulin injectable agents | 21 | 22 | 43
  Oral agents | 45 | 48 | 93

OUTCOME MEASURES:

1. Primary Outcome: Postprandial Glucose Control
Description: Percent of time spent in the glycemic target range of 100-180 mg/dL in the 4 hour postprandial period will be assessed using a continuous glucose monitoring (CGM) system.
Time Frame: 3 days
Population: A total of 110 participants received at least 4 meal boluses and had adequate 4-hr CG data for analysis. Results presented as percentage time in range 100-180 mg/dL in the 4 hour postprandial period for each group
Measure: Mean (Standard Deviation); unit: percentage of time in range (TIR)
Arm/Group | Group 1 Insulin Glargine and Novolog | Group 2 Insulin Glargine and Fiasp
Number analyzed (Participants) | 57 | 53
percentage of time in range (TIR) | 36.18 (29.78) | 45.22 (32.63)

2. Secondary Outcome: Glycemic Control While Hospitalized
Description: Percent of time spent in the glycemic target range of 100-180 mg/dL during the duration of the study will be assessed using a continuous glucose monitoring (CGM) system.
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: percentage of time in range (TIR)
Arm/Group | Group 1 Insulin Glargine and Novolog | Group 2 Insulin Glargine and Fiasp
Number analyzed (Participants) | 61 | 61
percentage of time in range (TIR) | 34.9 (26.0) | 39.9 (26.6)

3. Secondary Outcome: Percent of Time Spent in Glycemic Range of 70-140 mg/dL
Description: Percent of time spent in the glycemic target range of 70-140 mg/dL during the duration of the study assessed using a continuous glucose monitoring (CGM) system.
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: percentage of time in range (TIR)
Arm/Group | Group 1 Insulin Glargine and Novolog | Group 2 Insulin Glargine and Fiasp
Number analyzed (Participants) | 61 | 61
percentage of time in range (TIR) | 16.9 (18.4) | 20.2 (21.3)

4. Secondary Outcome: Percent of Time Spent With Hypoglycemia During Hospitalization
Description: The percent of time in three categories of hypoglycemia : <70 mg/dL, <54 mg/dL, and <40 mg/dL will be assessed using a CGM during hospitalization.
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: percentage of time in range (TIR)
Arm/Group | Group 1 Insulin Glargine and Novolog | Group 2 Insulin Glargine and Fiasp
Number analyzed (Participants) | 61 | 61
percentage of time in range (TIR)
  BG <70 dL/mg | 0.80 (2.1) | 1.52 (4.6)
  BG <54 dL/mg | 0.16 (0.6) | 0.53 (1.7)
  BG <40 dL/mg | 0.02 (0.08) | 0.10 (0.44)

5. Secondary Outcome: Percent of Nocturnal Time in Glycemic Target Range 100-180 mg/dL
Description: The percent of nocturnal time (from 00.01 AM to 5:59 AM) in the glycemic target range of 100-180 mg/dL
Time Frame: 3 days
Population: Only participants with 95% valid CGM data were included in this overnight analysis. This was a total of 108 participants- 56 in the Novolog group and 52 in the Fiasp group.
Measure: Mean (Standard Deviation); unit: percentage of time in range (TIR)
Arm/Group | Group 1 Insulin Glargine and Novolog | Group 2 Insulin Glargine and Fiasp
Number analyzed (Participants) | 56 | 52
percentage of time in range (TIR) | 36.7 (37.4) | 42.1 (40.7)

6. Secondary Outcome: Percent of Nocturnal Time Spent With Hypoglycemia
Description: The percent of nocturnal time (from 00.01 AM to 5:59 AM) in three categories of hypoglycemia: <70 mg/dL, <54 mg/dL, and <40 mg/dL will be assessed using CGM.
Time Frame: 3 days
Population: Patients with adequate overnight CGM data for analysis
Measure: Mean (Standard Deviation); unit: percent time in range
Arm/Group | Group 1 Insulin Glargine and Novolog | Group 2 Insulin Glargine and Fiasp
Number analyzed (Participants) | 56 | 52
percent time in range
  <70 mg/dL | 0.52 (2.44) | 1.12 (4.85)
  <54 mg/dL | 0.043 (0.24) | 0.22 (1.31)
  <40 | 0 (0) | 0.073 (0.56)

7. Secondary Outcome: Percent of Postprandial Time Spent With Level 1 Hyperglycemia
Description: The percent of time spent in level 1 hyperglycemia (181-239 mg/dL) will be assessed using CGM in the 4 hour postprandial period.
Time Frame: 4 hours postprandial
Population: There were 110 participants (57 in the Novolog arm and 53 in the Fiasp arm) with 4-hour postprandial data available for analysis
Measure: Mean (Standard Deviation); unit: percentage of time in range (TIR)
Arm/Group | Group 1 Insulin Glargine and Novolog | Group 2 Insulin Glargine and Fiasp
Number analyzed (Participants) | 57 | 53
percentage of time in range (TIR) | 30.1 (16.9) | 23.3 (19.2)

8. Secondary Outcome: Percent of Postprandial Time Spent With Level 2 Hyperglycemia
Description: The percent of time spent in level 2 hyperglycemia (>240 mg/dL) will be assessed using CGM in the 4 hour postprandial period.
Time Frame: 4 hours postprandial
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of time in range (TIR)
Arm/Group | Group 1 Insulin Glargine and Novolog | Group 2 Insulin Glargine and Fiasp
Number analyzed (Participants) | 57 | 53
percentage of time in range (TIR) | 30.3 (31.2) | 26.7 (31.2)

9. Secondary Outcome: Percent of Postprandial Time Spent With Hypoglycemia
Description: The percent of postprandial time in three categories of hypoglycemia will be assessed: <70 mg/dL, <54 mg/dL, and <40 mg/dL.
Time Frame: 4 hours postprandial
Measure: Mean (Standard Deviation); unit: percentage of time in range (TIR)
Arm/Group | Group 1 Insulin Glargine and Novolog | Group 2 Insulin Glargine and Fiasp
Number analyzed (Participants) | 57 | 53
percentage of time in range (TIR)
  BG <70 mg/dL | 0.70 (2.32) | 0.76 (3.37)
  BG <54 mg/dL | 0.14 (0.85) | 012 (0.75)
  BG <40 mg/dL | 0.01 (0.07) | 0.03 (0.19)

ADVERSE EVENTS:
Time Frame: During subject participation, on average 3 days
Description: Collected during the study
Arm/Group | Group 1 Insulin Glargine and Novolog | Group 2 Insulin Glargine and Fiasp
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/61 | 1/61
Other Adverse Events (participants affected / at risk) | 0/61 | 1/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Insulin Glargine and Novolog (N=61) | Group 2 Insulin Glargine and Fiasp (N=61)
transfer to higher level of care (General disorders) | 0 (0) | 1 (1) — After enrollment but before receiving any study medication pt became clinically worse and was transferred to a higher level of care. Subject was immediately discontinued from the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Insulin Glargine and Novolog (N=61) | Group 2 Insulin Glargine and Fiasp (N=61)
bleeding at CGM site (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — pt experienced bleeding at CGM site, sensor was removed and subject was discontinued from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT04460326/Prot_SAP_000.pdf